CLINICAL TRIAL: NCT02420561
Title: Motivational Interviewing to Reduce Substance Use Among Depression Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Foundation Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-03323
Record Dates: First submitted 2015-04-07; First posted 2015-04-20 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Depression; Substance-Related Disorders
Keywords: Depression; Substance-Related Disorders; Mental Health
MeSH Terms: conditions — Depression; Substance-Related Disorders; Psychological Well-Being | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing (Experimental): The motivational interviewing (MI) intervention consisted of one 45-minute in-person MI session followed by two 15-minute telephone "booster" sessions
  Interventions: Behavioral: Motivational Interviewing
- Control (Active Comparator): Participants received a brochure on alcohol and drug use risks.
  Interventions: Behavioral: Control (brochure)

INTERVENTIONS:
Behavioral: Motivational Interviewing — * One in-person motivational interviewing session intervention that lasts for 45-minutes
  * Additional two 15-minute telephone "booster" sessions post in-person 45 minute sessions
  Arms: Motivational Interviewing
Behavioral: Control (brochure) — Participants received a brochure on alcohol and drug use risks.
  Arms: Control

SUMMARY:
The study aims to evaluate the effectiveness of an intervention to reduce alcohol and drug use and depression symptoms, improve functional status and promote appropriate health services utilization, in a sample of 300 adults seeking treatment for depression who also report hazardous drinking or drug use with depression.

DETAILED DESCRIPTION:
This study addresses important questions regarding how to identify and treat patients in Psychiatry who present for services with alcohol or drug use that may exacerbate depression. The investigators propose a study of Brief Motivational Intervention (BMI) to reduce drug and alcohol use among patients with depression, and to enhance engagement with a Kaiser Chemical Dependency Recovery Program (CDRP) as needed. Patients with depression who use drugs or alcohol even at sub-diagnostic levels are at high risk for escalation of substance problems. BMI is an innovative, evidence-based approach that could decrease drug and alcohol use and improve outcomes. But it has not been tested among depression patients. This study sample will include 300 outpatients in treatment for depression in Kaiser Permanente Northern California Hayward/Fremont Psychiatry. Inclusion criteria are based on drug use (any illicit drug use and non-prescribed use of prescription drugs) and hazardous drinking (i.e., ≥ 3 drinks in a day for women and ≥ 4 drinks in a day for men), and moderate to severe depression symptoms at intake. Three hundred patients will be randomized to receive one in-person BMI session and two telephone BMI sessions within 6 weeks of intake (intervention) or a brochure on risks of drug and alcohol use (control). The investigators anticipate that the intervention will be effective in reducing frequency of drug use and hazardous drinking at 3-, 6-, and 12-month telephone follow-up interviews; improving mood and functional outcomes; increasing depression treatment retention (number of psychiatry visits, based on Healthcare Effectiveness Data and Information Set (HEDIS) standards); and facilitating patient initiation of chemical dependency program treatment if needed, and will be cost effective. For the improvement of patient care, it will also yield important information on integrating alcohol and drug intervention in Psychiatry and how best to help patients access specialty CDRP services when needed.

ELIGIBILITY:
Inclusion Criteria:

* Hazardous drinking (i.e., ≥ 3 drinks in a day for women and ≥ 4 drinks in a day for men)
* Drug use (including any illicit drug use and non-prescribed use of prescription drugs in the prior 30 days)
* Moderate or greater symptoms of depression based on a score of ≥ 5 on the Patient Health Questionnaire (PHQ-9)

Exclusion Criteria:

* Current mania or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Hazardous drinking in the prior 30 days (Self-reported number of days of hazardous drinking) | 6 months
  Self-reported number of days of hazardous drinking (3+ drinks per day for women / 4+ drinks per day for men) in the prior 30 days.
Drug use in the prior 30 days (Self-reported number of days of drug use) | 6 months
  Self-reported number of days of drug use (illegal drug use or misuse of prescription drugs) in the 30 prior days.
Hazardous drinking in the prior 30 days (Self-reported number of days of hazardous drinking) | 12 months
  Self-reported number of days of hazardous drinking (3+ drinks per day for women / 4+ drinks per day for men) in the prior 30 days. We examine the change between use at 6 months and use at 12 months to measure long term intervention impact.
Drug use in the prior 30 days (Self-reported number of days of drug use) | 12 months
  Self-reported number of days of drug use (illegal drug use or misuse of prescription drugs) in the 30 prior days. We examine the change in use between 6 months and 12 months to measure long term intervention impact.

SECONDARY OUTCOMES:
Depression symptoms (Patient health questionnaire (PHQ-9) score) | 12 months
  measured at follow up telephone interviews.The PHQ-9 assesses frequency of 9 types of problems over the past 2 weeks; answers range from 0 (not at all) to 3 (nearly every day). If at least 4 of 9 are >0, the sum of item scores is used to indicate severity of depression: 1-4 Minimal; 5-9 Mild; 10-14 Moderate; 15-19 Moderately Severe; 20-27 Severe.
Adequate mental health treatment (Number of participants receiving 12 weeks' continuous treatment at the Kaiser Permanente Outpatient Psychiatry Department) | 3 months
  Number of participants receiving 12 weeks' continuous treatment at the Kaiser Permanente Outpatient Psychiatry Department

CONTACTS AND LOCATIONS:
Overall Officials: Derek D Satre, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Permanente Medical Center Southern Alameda County, Union City, California, United States

REFERENCES:
- [Background] Babor TF, McRee BG, Kassebaum PA, Grimaldi PL, Ahmed K, Bray J. Screening, Brief Intervention, and Referral to Treatment (SBIRT): toward a public health approach to the management of substance abuse. Subst Abus. 2007;28(3):7-30. doi: 10.1300/J465v28n03_03. PMID 18077300
- [Background] Madras BK, Compton WM, Avula D, Stegbauer T, Stein JB, Clark HW. Screening, brief interventions, referral to treatment (SBIRT) for illicit drug and alcohol use at multiple healthcare sites: comparison at intake and 6 months later. Drug Alcohol Depend. 2009 Jan 1;99(1-3):280-95. doi: 10.1016/j.drugalcdep.2008.08.003. Epub 2008 Oct 16. PMID 18929451
- [Background] Substance Abuse and Mental Health Services Administration, Center for Substance Abuse Treatment. Screening, brief intervention, and referral to treatment. What is SBIRT? . http://sbirt.samhsa.gov/index.htm. Published 2008. Accessed September 1, 2009
- [Background] Carroll KM, Ball SA, Nich C, Martino S, Frankforter TL, Farentinos C, Kunkel LE, Mikulich-Gilbertson SK, Morgenstern J, Obert JL, Polcin D, Snead N, Woody GE; National Institute on Drug Abuse Clinical Trials Network. Motivational interviewing to improve treatment engagement and outcome in individuals seeking treatment for substance abuse: a multisite effectiveness study. Drug Alcohol Depend. 2006 Feb 28;81(3):301-12. doi: 10.1016/j.drugalcdep.2005.08.002. Epub 2005 Sep 28. PMID 16169159
- [Background] Carroll KM, Libby B, Sheehan J, Hyland N. Motivational interviewing to enhance treatment initiation in substance abusers: an effectiveness study. Am J Addict. 2001 Fall;10(4):335-9. doi: 10.1080/aja.10.4.335.339. PMID 11783748
- [Background] Dunn C, Deroo L, Rivara FP. The use of brief interventions adapted from motivational interviewing across behavioral domains: a systematic review. Addiction. 2001 Dec;96(12):1725-42. doi: 10.1046/j.1360-0443.2001.961217253.x. PMID 11784466
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision. Washington, DC: American Psychiatric Association, 2000.
- [Background] McCabe SE, West BT, Morales M, Cranford JA, Boyd CJ. Does early onset of non-medical use of prescription drugs predict subsequent prescription drug abuse and dependence? Results from a national study. Addiction. 2007 Dec;102(12):1920-30. doi: 10.1111/j.1360-0443.2007.02015.x. Epub 2007 Oct 4. PMID 17916222
- [Background] Zahradnik A, Otto C, Crackau B, Lohrmann I, Bischof G, John U, Rumpf HJ. Randomized controlled trial of a brief intervention for problematic prescription drug use in non-treatment-seeking patients. Addiction. 2009 Jan;104(1):109-17. doi: 10.1111/j.1360-0443.2008.02421.x. PMID 19133895
- [Background] Weingartner K, Robison J, Fogel D, Gruman C. Depression and substance use in a middle aged and older Puerto Rican population. J Cross Cult Gerontol. 2002;17(2):173-93. doi: 10.1023/a:1015861002809. PMID 14617972
- [Background] Compton WM, Volkow ND. Abuse of prescription drugs and the risk of addiction. Drug Alcohol Depend. 2006 Jun;83 Suppl 1:S4-7. doi: 10.1016/j.drugalcdep.2005.10.020. Epub 2006 Mar 23. PMID 16563663
- [Background] Weisner C, McLellan AT, Hunkeler EM. Addiction severity index data from general membership and treatment samples of HMO members. One case of norming the ASI. J Subst Abuse Treat. 2000 Sep;19(2):103-9. doi: 10.1016/s0740-5472(99)00103-8. PMID 10963921
- [Background] Braden JB, Sullivan MD, Ray GT, Saunders K, Merrill J, Silverberg MJ, Rutter CM, Weisner C, Banta-Green C, Campbell C, Von Korff M. Trends in long-term opioid therapy for noncancer pain among persons with a history of depression. Gen Hosp Psychiatry. 2009 Nov-Dec;31(6):564-70. doi: 10.1016/j.genhosppsych.2009.07.003. Epub 2009 Aug 27. PMID 19892215
- [Background] Weisner CM, Campbell CI, Ray TG, Saunders K, Merrill JO, Banta-Green C, Sullivan MD, Silverberg MJ, Mertens JR, Boudreau D, Von Korff M. Trends in prescribed opioid therapy for non-cancer pain for individuals with prior substance use disorders. Pain. 2009 Oct;145(3):287-293. doi: 10.1016/j.pain.2009.05.006. Epub 2009 Jul 5. PMID 19581051
- [Background] National Institute on Drug Abuse. NM Assist: Screening for drug use in general medical settings. http://ww1.drugabuse.gov/nmassist/. Published 2009. Updated Sep 17, 2009. Accessed Oct 8, 2009
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Lu Y. Integrating primary medical care with addiction treatment: a randomized controlled trial. JAMA. 2001 Oct 10;286(14):1715-23. doi: 10.1001/jama.286.14.1715. PMID 11594896
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Hunkeler EM, Hu T, Selby JV. The outcome and cost of alcohol and drug treatment in an HMO: day hospital versus traditional outpatient regimens. Health Serv Res. 2000 Oct;35(4):791-812. PMID 11055449
- [Background] Compton PA, Wu SM, Schieffer B, Pham Q, Naliboff BD. Introduction of a self-report version of the Prescription Drug Use Questionnaire and relationship to medication agreement noncompliance. J Pain Symptom Manage. 2008 Oct;36(4):383-95. doi: 10.1016/j.jpainsymman.2007.11.006. Epub 2008 Jun 3. PMID 18508231
- [Background] Butler SF, Budman SH, Fernandez KC, Houle B, Benoit C, Katz N, Jamison RN. Development and validation of the Current Opioid Misuse Measure. Pain. 2007 Jul;130(1-2):144-56. doi: 10.1016/j.pain.2007.01.014. Epub 2007 May 9. PMID 17493754
- [Background] Hepner KA, Hunter SB, Edelen MO, Zhou AJ, Watkins K. A comparison of two depressive symptomatology measures in residential substance abuse treatment clients. J Subst Abuse Treat. 2009 Oct;37(3):318-25. doi: 10.1016/j.jsat.2009.03.005. Epub 2009 Apr 8. PMID 19359127
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Manwell LB, Fleming MF, Mundt MP, Stauffacher EA, Barry KL. Treatment of problem alcohol use in women of childbearing age: results of a brief intervention trial. Alcohol Clin Exp Res. 2000 Oct;24(10):1517-24. PMID 11045860
- [Background] Rickles NM, Svarstad BL. Relationships between multiple self-reported nonadherence measures and pharmacy records. Res Social Adm Pharm. 2007 Dec;3(4):363-77. doi: 10.1016/j.sapharm.2006.11.001. PMID 18082873
- [Background] Satre D, Wolfe W, Eisendrath S, Weisner C. Computerized screening for alcohol and drug use among adults seeking outpatient psychiatric services. Psychiatr Serv. 2008 Apr;59(4):441-4. doi: 10.1176/ps.2008.59.4.441. PMID 18378846
- [Background] Roeloffs CA, Fink A, Unutzer J, Tang L, Wells KB. Problematic substance use, depressive symptoms, and gender in primary care. Psychiatr Serv. 2001 Sep;52(9):1251-3. doi: 10.1176/appi.ps.52.9.1251. PMID 11533403
- [Background] Kessler RC. The epidemiology of dual diagnosis. Biol Psychiatry. 2004 Nov 15;56(10):730-7. doi: 10.1016/j.biopsych.2004.06.034. PMID 15556117
- [Background] Sullivan LE, Fiellin DA, O'Connor PG. The prevalence and impact of alcohol problems in major depression: a systematic review. Am J Med. 2005 Apr;118(4):330-41. doi: 10.1016/j.amjmed.2005.01.007. PMID 15808128
- [Background] Agosti V, Nunes E, Levin F. Rates of psychiatric comorbidity among U.S. residents with lifetime cannabis dependence. Am J Drug Alcohol Abuse. 2002 Nov;28(4):643-52. doi: 10.1081/ada-120015873. PMID 12492261
- [Background] Wisniewski SR, Fava M, Trivedi MH, Thase ME, Warden D, Niederehe G, Friedman ES, Biggs MM, Sackeim HA, Shores-Wilson K, McGrath PJ, Lavori PW, Miyahara S, Rush AJ. Acceptability of second-step treatments to depressed outpatients: a STAR*D report. Am J Psychiatry. 2007 May;164(5):753-60. doi: 10.1176/ajp.2007.164.5.753. PMID 17475734
- [Background] Worthington J, Fava M, Agustin C, Alpert J, Nierenberg AA, Pava JA, Rosenbaum JF. Consumption of alcohol, nicotine, and caffeine among depressed outpatients. Relationship with response to treatment. Psychosomatics. 1996 Nov-Dec;37(6):518-22. doi: 10.1016/S0033-3182(96)71515-3. PMID 8942202
- [Background] Kuo PH, Gardner CO, Kendler KS, Prescott CA. The temporal relationship of the onsets of alcohol dependence and major depression: using a genetically informative study design. Psychol Med. 2006 Aug;36(8):1153-62. doi: 10.1017/S0033291706007860. Epub 2006 May 31. PMID 16734951
- [Background] Dixit AR, Crum RM. Prospective study of depression and the risk of heavy alcohol use in women. Am J Psychiatry. 2000 May;157(5):751-8. doi: 10.1176/appi.ajp.157.5.751. PMID 10784468
- [Background] Weisner C, Matzger H. Missed opportunities in addressing drinking behavior in medical and mental health services. Alcohol Clin Exp Res. 2003 Jul;27(7):1132-41. doi: 10.1097/01.ALC.0000075546.38349.69. PMID 12878919
- [Background] Abraham HD, Fava M. Order of onset of substance abuse and depression in a sample of depressed outpatients. Compr Psychiatry. 1999 Jan-Feb;40(1):44-50. doi: 10.1016/s0010-440x(99)90076-7. PMID 9924877
- [Background] Satre DD, Wolfe W, Eisendrath S, et al. Alcohol and drug use in outpatient mental health: prevalence, motivation to reduce drinking, and impact on treatment retention. Annual meeting of the American Psychological Association, San Francisco, CA, Aug 19, 2007
- [Background] Merikangas KR, Ames M, Cui L, Stang PE, Ustun TB, Von Korff M, Kessler RC. The impact of comorbidity of mental and physical conditions on role disability in the US adult household population. Arch Gen Psychiatry. 2007 Oct;64(10):1180-8. doi: 10.1001/archpsyc.64.10.1180. PMID 17909130
- [Background] Goetzel RZ, Hawkins K, Ozminkowski RJ, Wang S. The health and productivity cost burden of the "top 10" physical and mental health conditions affecting six large U.S. employers in 1999. J Occup Environ Med. 2003 Jan;45(1):5-14. doi: 10.1097/00043764-200301000-00007. PMID 12553174
- [Background] Wang PS, Simon G, Kessler RC. The economic burden of depression and the cost-effectiveness of treatment. Int J Methods Psychiatr Res. 2003;12(1):22-33. doi: 10.1002/mpr.139. PMID 12830307
- [Background] National Institute on Alcohol Abuse and Alcoholism. Helping patients who drink too much: a clinician's guide, updated 2005 edition. Rockville, MD: National Institute on Alcohol Abuse and Alcoholism; 2005: http://pubs.niaaa.nih.gov/publications/Practitioner/CliniciansGuide2005/clinicians_guide.htm. Updated 2007 Jan. Accessed Jul
- [Background] Adamson SJ, Sellman JD. Five-year outcomes of alcohol-dependent persons treated with motivational enhancement. J Stud Alcohol Drugs. 2008 Jul;69(4):589-93. doi: 10.15288/jsad.2008.69.589. PMID 18612575
- [Background] Lang E, Engelander M, Brooke T. Report of an integrated brief intervention with self-defined problem cannabis users. J Subst Abuse Treat. 2000 Sep;19(2):111-6. doi: 10.1016/s0740-5472(99)00104-x. PMID 10963922
- [Background] Miller WR, Yahne CE, Tonigan JS. Motivational interviewing in drug abuse services: a randomized trial. J Consult Clin Psychol. 2003 Aug;71(4):754-63. doi: 10.1037/0022-006x.71.4.754. PMID 12924680
- [Background] Carroll KM. Behavioral therapies for co-occurring substance use and mood disorders. Biol Psychiatry. 2004 Nov 15;56(10):778-84. doi: 10.1016/j.biopsych.2004.07.010. PMID 15556123
- [Background] Kessler RC. Epidemiology of women and depression. J Affect Disord. 2003 Mar;74(1):5-13. doi: 10.1016/s0165-0327(02)00426-3. PMID 12646294
- [Background] Culbertson FM. Depression and gender. An international review. Am Psychol. 1997 Jan;52(1):25-31. doi: 10.1037//0003-066x.52.1.25. PMID 9017929
- [Background] Helzer JE, Bucholz K, Robins LN. Five communities in the United States: results of the Epidemiologic Catchment Area study. In: Helzer JE, Canino GJ, eds. Alcoholism in North American, Europe, and Asia. New York: Oxford University Press, 1992:71-95
- [Background] Farrell M. Cannabis dependence and withdrawal. Addiction. 1999 Sep;94(9):1277-8. doi: 10.1046/j.1360-0443.1999.94912771.x. No abstract available. PMID 10615714
- [Background] Substance Abuse and Mental Health Services Administration. National Household Survey on Drug Abuse: Population Estimates 1998. Vol H-11. Rockville, MD: Department of Health and Human Services, Office of Applied Studies, 1999
- [Background] Katerndahl DA, Realini JP. Relationship between substance abuse and panic attacks. Addict Behav. 1999 Sep-Oct;24(5):731-6. doi: 10.1016/s0306-4603(98)00078-1. PMID 10574314
- [Background] Sbrana A, Bizzarri JV, Rucci P, Gonnelli C, Doria MR, Spagnolli S, Ravani L, Raimondi F, Dell'Osso L, Cassano GB. The spectrum of substance use in mood and anxiety disorders. Compr Psychiatry. 2005 Jan-Feb;46(1):6-13. doi: 10.1016/j.comppsych.2004.07.017. PMID 15714188
- [Background] Dannon PN, Lowengrub K, Amiaz R, Grunhaus L, Kotler M. Comorbid cannabis use and panic disorder: short term and long term follow-up study. Hum Psychopharmacol. 2004 Mar;19(2):97-101. doi: 10.1002/hup.560. PMID 14994319
- [Background] Bovasso GB. Cannabis abuse as a risk factor for depressive symptoms. Am J Psychiatry. 2001 Dec;158(12):2033-7. doi: 10.1176/appi.ajp.158.12.2033. PMID 11729021
- [Background] Rey JM, Martin A, Krabman P. Is the party over? Cannabis and juvenile psychiatric disorder: the past 10 years. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1194-205. doi: 10.1097/01.chi.0000135623.12843.60. PMID 15381886
- [Background] Chen CY, Wagner FA, Anthony JC. Marijuana use and the risk of Major Depressive Episode. Epidemiological evidence from the United States National Comorbidity Survey. Soc Psychiatry Psychiatr Epidemiol. 2002 May;37(5):199-206. doi: 10.1007/s00127-002-0541-z. PMID 12107710
- [Background] Lynskey MT, Glowinski AL, Todorov AA, Bucholz KK, Madden PA, Nelson EC, Statham DJ, Martin NG, Heath AC. Major depressive disorder, suicidal ideation, and suicide attempt in twins discordant for cannabis dependence and early-onset cannabis use. Arch Gen Psychiatry. 2004 Oct;61(10):1026-32. doi: 10.1001/archpsyc.61.10.1026. PMID 15466676
- [Background] Barry KL, Milner K, Blow FC, Impens A, Welsh D, Amash J. Screening psychiatric emergency department patients with major mental illnesses for at-risk drinking. Psychiatr Serv. 2006 Jul;57(7):1039-42. doi: 10.1176/ps.2006.57.7.1039. PMID 16816292
- [Background] Akincigil A, Bowblis JR, Levin C, Walkup JT, Jan S, Crystal S. Adherence to antidepressant treatment among privately insured patients diagnosed with depression. Med Care. 2007 Apr;45(4):363-9. doi: 10.1097/01.mlr.0000254574.23418.f6. PMID 17496721
- [Background] National Cannabis Prevention and Information Centre (NCPIC). Cannabis and prescribed medications. http://ncpic.org.au/ncpic/publications/factsheets/article/cannabis-and-prescribed-medications;. Published 2008. Accessed Sep 28, 2009
- [Background] Wilens TE, Biederman J, Spencer TJ. Case study: adverse effects of smoking marijuana while receiving tricyclic antidepressants. J Am Acad Child Adolesc Psychiatry. 1997 Jan;36(1):45-8. doi: 10.1097/00004583-199701000-00016. PMID 9000780
- [Background] O'Dell LE, George FR, Ritz MC. Antidepressant drugs appear to enhance cocaine-induced toxicity. Exp Clin Psychopharmacol. 2000 Feb;8(1):133-41. doi: 10.1037//1064-1297.8.1.133. PMID 10743914
- [Background] Stein MD, Herman DS, Solomon DA, Anthony JL, Anderson BJ, Ramsey SE, Miller IW. Adherence to treatment of depression in active injection drug users: the minerva study. J Subst Abuse Treat. 2004 Mar;26(2):87-93. doi: 10.1016/S0740-5472(03)00160-0. PMID 15050085
- [Background] National Institute on Drug Abuse. Depression elevates suicide risk in substance-abusing adolescents. NIDA Notes. 2005;19(6). http://www.drugabuse.gov/NIDA_notes/NNvol19N6/Depression.html. Accessed Oct 15, 2009.
- [Background] National Institute of Mental Health. Depression. http://www.nimh.nih.gov/publicat/depression.cfm. Published 2000. Updated 2006 Sep 13. Accessed 2007 Jan 8
- [Background] National Institute of Mental Health. Medications. http://www.nimh.nih.gov/health/publications/medications/complete-publication.shtml#pub8. Published 2008. Accessed Oct 15, 2009.
- [Background] Fleming MF, Manwell LB, Barry KL, Johnson K. At-risk drinking in an HMO primary care sample: prevalence and health policy implications. Am J Public Health. 1998 Jan;88(1):90-3. doi: 10.2105/ajph.88.1.90. PMID 9584040
- [Background] Dawson DA, Grant BF, Chou SP, Pickering RP. Subgroup variation in U.S. drinking patterns: results of the 1992 national longitudinal alcohol epidemiologic study. J Subst Abuse. 1995;7(3):331-44. doi: 10.1016/0899-3289(95)90026-8. PMID 8749792
- [Background] Archer L, Grant BF, Dawson DA. What if Americans drank less? The potential effect on the prevalence of alcohol abuse and dependence. Am J Public Health. 1995 Jan;85(1):61-6. doi: 10.2105/ajph.85.1.61. PMID 7832263
- [Background] Grant BF. Comorbidity between DSM-IV drug use disorders and major depression: results of a national survey of adults. J Subst Abuse. 1995;7(4):481-97. doi: 10.1016/0899-3289(95)90017-9. PMID 8838629
- [Background] Graham K, Massak A, Demers A, Rehm J. Does the association between alcohol consumption and depression depend on how they are measured? Alcohol Clin Exp Res. 2007 Jan;31(1):78-88. doi: 10.1111/j.1530-0277.2006.00274.x. PMID 17207105
- [Background] O'Donnell K, Wardle J, Dantzer C, Steptoe A. Alcohol consumption and symptoms of depression in young adults from 20 countries. J Stud Alcohol. 2006 Nov;67(6):837-40. doi: 10.15288/jsa.2006.67.837. PMID 17061000
- [Background] Alati R, Lawlor DA, Mamun AA, Williams GM, Najman JM, O'Callaghan M, Bor W. Is there a fetal origin of depression? Evidence from the Mater University Study of Pregnancy and its outcomes. Am J Epidemiol. 2007 Mar 1;165(5):575-82. doi: 10.1093/aje/kwk036. Epub 2006 Dec 5. PMID 17148497
- [Background] Rodgers B, Korten AE, Jorm AF, Jacomb PA, Christensen H, Henderson AS. Non-linear relationships in associations of depression and anxiety with alcohol use. Psychol Med. 2000 Mar;30(2):421-32. doi: 10.1017/s0033291799001865. PMID 10824662
- [Background] Midanik LT, Tam TW, Weisner C. Concurrent and simultaneous drug and alcohol use: results of the 2000 National Alcohol Survey. Drug Alcohol Depend. 2007 Sep 6;90(1):72-80. doi: 10.1016/j.drugalcdep.2007.02.024. Epub 2007 Apr 18. PMID 17446013
- [Background] Davis LL, Rush JA, Wisniewski SR, Rice K, Cassano P, Jewell ME, Biggs MM, Shores-Wilson K, Balasubramani GK, Husain MM, Quitkin FM, McGrath PJ. Substance use disorder comorbidity in major depressive disorder: an exploratory analysis of the Sequenced Treatment Alternatives to Relieve Depression cohort. Compr Psychiatry. 2005 Mar-Apr;46(2):81-9. doi: 10.1016/j.comppsych.2004.07.025. PMID 15723023
- [Background] Sanderson WC, Beck AT, Beck J. Syndrome comorbidity in patients with major depression or dysthymia: prevalence and temporal relationships. Am J Psychiatry. 1990 Aug;147(8):1025-8. doi: 10.1176/ajp.147.8.1025. PMID 2375436
- [Background] McDermut W, Mattia J, Zimmerman M. Comorbidity burden and its impact on psychosocial morbidity in depressed outpatients. J Affect Disord. 2001 Aug;65(3):289-95. doi: 10.1016/s0165-0327(00)00220-2. PMID 11511409
- [Background] Fava M, Abraham M, Alpert J, Nierenberg AA, Pava JA, Rosenbaum JF. Gender differences in Axis I comorbidity among depressed outpatients. J Affect Disord. 1996 Jun 5;38(2-3):129-33. doi: 10.1016/0165-0327(96)00004-3. PMID 8791181
- [Background] Gratzer D, Levitan RD, Sheldon T, Toneatto T, Rector NA, Goering P. Lifetime rates of alcoholism in adults with anxiety, depression, or co-morbid depression/anxiety: a community survey of Ontario. J Affect Disord. 2004 Apr;79(1-3):209-15. doi: 10.1016/S0165-0327(02)00355-5. PMID 15023496
- [Background] Smith SM, Stinson FS, Dawson DA, Goldstein R, Huang B, Grant BF. Race/ethnic differences in the prevalence and co-occurrence of substance use disorders and independent mood and anxiety disorders: Results from the National Epidemiologic Survey on Alcohol and Related Conditions. Psychol Med. 2006 Jul;36(7):987-98. doi: 10.1017/S0033291706007690. Epub 2006 May 2. PMID 16650344
- [Background] Scott J, Gilvarry E, Farrell M. Managing anxiety and depression in alcohol and drug dependence. Addict Behav. 1998 Nov-Dec;23(6):919-31. doi: 10.1016/s0306-4603(98)00074-4. PMID 9801726
- [Background] Institute of Medicine (US) Committee on Quality Assurance and Accreditation Guidelines for Managed Behavioral Health Care; Edmunds M, Frank R, Hogan M, McCarty D, Robinson-Beale R, Weisner C, editors. Managing Managed Care: Quality Improvement in Behavioral Health. Washington (DC): National Academies Press (US); 1997. Available from http://www.ncbi.nlm.nih.gov/books/NBK233228/ PMID 25121327
- [Background] Rounsaville BJ, Petry NM, Carroll KM. Single versus multiple drug focus in substance abuse clinical trials research. Drug Alcohol Depend. 2003 May 21;70(2):117-25. doi: 10.1016/s0376-8716(03)00033-4. PMID 12732403
- [Background] Martin CS, Kaczynski NA, Maisto SA, Tarter RE. Polydrug use in adolescent drinkers with and without DSM-IV alcohol abuse and dependence. Alcohol Clin Exp Res. 1996 Sep;20(6):1099-1108. doi: 10.1111/j.1530-0277.1996.tb01953.x. PMID 8892534
- [Background] Ross HE. Benzodiazepine use and anxiolytic abuse and dependence in treated alcoholics. Addiction. 1993 Feb;88(2):209-18. doi: 10.1111/j.1360-0443.1993.tb00804.x. PMID 8106063
- [Background] Gossop M, Manning V, Ridge G. Concurrent use and order of use of cocaine and alcohol: behavioural differences between users of crack cocaine and cocaine powder. Addiction. 2006 Sep;101(9):1292-8. doi: 10.1111/j.1360-0443.2006.01497.x. PMID 16911728
- [Background] Caetano R, Weisner C. The association between DSM-III-R alcohol dependence, psychological distress and drug use. Addiction. 1995 Mar;90(3):351-9. doi: 10.1046/j.1360-0443.1995.9033515.x. PMID 7735020
- [Background] Zayas LH, Rojas M, Malgady RG. Alcohol and drug use, and depression among Hispanic men in early adulthood. Am J Community Psychol. 1998 Jun;26(3):425-38. doi: 10.1023/a:1022111221380. PMID 9726116
- [Background] Brunette MF, Noordsy DL, Xie H, Drake RE. Benzodiazepine use and abuse among patients with severe mental illness and co-occurring substance use disorders. Psychiatr Serv. 2003 Oct;54(10):1395-401. doi: 10.1176/appi.ps.54.10.1395. PMID 14557527
- [Background] Brown RA, Monti PM, Myers MG, Martin RA, Rivinus T, Dubreuil ME, Rohsenow DJ. Depression among cocaine abusers in treatment: relation to cocaine and alcohol use and treatment outcome. Am J Psychiatry. 1998 Feb;155(2):220-5. doi: 10.1176/ajp.155.2.220. PMID 9464201
- [Background] Li TK, Hewitt BG, Grant BF. Alcohol use disorders and mood disorders: a National Institute on Alcohol Abuse and Alcoholism perspective. Biol Psychiatry. 2004 Nov 15;56(10):718-20. doi: 10.1016/j.biopsych.2004.03.006. No abstract available. PMID 15556112
- [Background] Degenhardt L, Hall W, Lynskey M. Exploring the association between cannabis use and depression. Addiction. 2003 Nov;98(11):1493-504. doi: 10.1046/j.1360-0443.2003.00437.x. PMID 14616175
- [Background] Bambico FR, Katz N, Debonnel G, Gobbi G. Cannabinoids elicit antidepressant-like behavior and activate serotonergic neurons through the medial prefrontal cortex. J Neurosci. 2007 Oct 24;27(43):11700-11. doi: 10.1523/JNEUROSCI.1636-07.2007. PMID 17959812
- [Background] Hayatbakhsh MR, Najman JM, Jamrozik K, Mamun AA, Alati R, Bor W. Cannabis and anxiety and depression in young adults: a large prospective study. J Am Acad Child Adolesc Psychiatry. 2007 Mar;46(3):408-417. doi: 10.1097/chi.0b013e31802dc54d. PMID 17314727
- [Background] Schinke SP, Fang L, Cole KC. Substance use among early adolescent girls: risk and protective factors. J Adolesc Health. 2008 Aug;43(2):191-4. doi: 10.1016/j.jadohealth.2007.12.014. Epub 2008 Apr 11. PMID 18639794
- [Background] Schepis TS, Krishnan-Sarin S. Characterizing adolescent prescription misusers: a population-based study. J Am Acad Child Adolesc Psychiatry. 2008 Jul;47(7):745-754. doi: 10.1097/CHI.0b013e318172ef0ld. PMID 18520963
- [Background] Herbeck DM, Hser YI, Lu AT, Stark ME, Paredes A. A 12-year follow-up study of psychiatric symptomatology among cocaine-dependent men. Addict Behav. 2006 Nov;31(11):1974-87. doi: 10.1016/j.addbeh.2006.01.013. Epub 2006 Feb 28. PMID 16503094
- [Background] Siqueland L, Horn A, Moras K, Woody G, Weiss R, Blaine J, Bishop S, Barber J, Thase M. Cocaine-induced mood disorder: prevalence rates and psychiatric symptoms in an outpatient cocaine-dependent sample. Am J Addict. 1999 Spring;8(2):165-9. doi: 10.1080/105504999305974. PMID 10365197
- [Background] Havassy BE, Arns PG. Relationship of cocaine and other substance dependence to well-being of high-risk psychiatric patients. Psychiatr Serv. 1998 Jul;49(7):935-40. doi: 10.1176/ps.49.7.935. PMID 9661229
- [Background] Rounsaville BJ. Treatment of cocaine dependence and depression. Biol Psychiatry. 2004 Nov 15;56(10):803-9. doi: 10.1016/j.biopsych.2004.05.009. PMID 15556126
- [Background] Conner KR, Pinquart M, Holbrook AP. Meta-analysis of depression and substance use and impairment among cocaine users. Drug Alcohol Depend. 2008 Nov 1;98(1-2):13-23. doi: 10.1016/j.drugalcdep.2008.05.005. Epub 2008 Jun 27. PMID 18585871
- [Background] Zweben JE, Cohen JB, Christian D, Galloway GP, Salinardi M, Parent D, Iguchi M; Methamphetamine Treatment Project. Psychiatric symptoms in methamphetamine users. Am J Addict. 2004 Mar-Apr;13(2):181-90. doi: 10.1080/10550490490436055. PMID 15204668
- [Background] Leamon MH, Canning RD, Benjamin L. The impact of amphetamine-related disorders on community psychiatric emergency services: 1993-1997. Am J Addict. 2000 Winter;9(1):70-8. doi: 10.1080/10550490050172245. PMID 10914295
- [Background] Castaneda R, Sussman N, Levy R, O'Malley M, Westreich L. A review of the effects of moderate alcohol intake on psychiatric and sleep disorders. Recent Dev Alcohol. 1998;14:197-226. doi: 10.1007/0-306-47148-5_9. PMID 9751947
- [Background] Cornelius JR, Salloum IM, Mezzich J, Cornelius MD, Fabrega H Jr, Ehler JG, Ulrich RF, Thase ME, Mann JJ. Disproportionate suicidality in patients with comorbid major depression and alcoholism. Am J Psychiatry. 1995 Mar;152(3):358-64. doi: 10.1176/ajp.152.3.358. PMID 7864260
- [Background] Salloum IM, Mezzich JE, Cornelius J, Day NL, Daley D, Kirisci L. Clinical profile of comorbid major depression and alcohol use disorders in an initial psychiatric evaluation. Compr Psychiatry. 1995 Jul-Aug;36(4):260-6. doi: 10.1016/s0010-440x(95)90070-5. PMID 7554869
- [Background] Waller SJ, Lyons JS, Costantini-Ferrando MF. Impact of comorbid affective and alcohol use disorders on suicidal ideation and attempts. J Clin Psychol. 1999 May;55(5):585-95. doi: 10.1002/(sici)1097-4679(199905)55:53.0.co;2-u. PMID 10392789
- [Background] Bolton J, Cox B, Clara I, Sareen J. Use of alcohol and drugs to self-medicate anxiety disorders in a nationally representative sample. J Nerv Ment Dis. 2006 Nov;194(11):818-25. doi: 10.1097/01.nmd.0000244481.63148.98. PMID 17102705
- [Background] Holahan CJ, Moos RH, Holahan CK, Cronkite RC, Randall PK. Drinking to cope and alcohol use and abuse in unipolar depression: a 10-year model. J Abnorm Psychol. 2003 Feb;112(1):159-65. PMID 12653424
- [Background] Nunes EV, Levin FR. Treatment of depression in patients with alcohol or other drug dependence: a meta-analysis. JAMA. 2004 Apr 21;291(15):1887-96. doi: 10.1001/jama.291.15.1887. PMID 15100209
- [Background] Anderson B. HEDIS antidepressant medication management measures and performance-based measures: an opportunity for improvement in depression care. Am J Manag Care. 2007 Nov;13(4 Suppl):S98-102. PMID 18041869
- [Background] Cantrell CR, Eaddy MT, Shah MB, Regan TS, Sokol MC. Methods for evaluating patient adherence to antidepressant therapy: a real-world comparison of adherence and economic outcomes. Med Care. 2006 Apr;44(4):300-3. doi: 10.1097/01.mlr.0000204287.82701.9b. PMID 16565629
- [Background] Bricker JB, Russo J, Stein MB, Sherbourne C, Craske M, Schraufnagel TJ, Roy-Byrne P. Does occasional cannabis use impact anxiety and depression treatment outcomes?: Results from a randomized effectiveness trial. Depress Anxiety. 2007;24(6):392-8. doi: 10.1002/da.20248. PMID 17096386
- [Background] Mueller MR, Shah NG, Landen MG. Unintentional prescription drug overdose deaths in New Mexico, 1994-2003. Am J Prev Med. 2006 May;30(5):423-9. doi: 10.1016/j.amepre.2005.12.011. PMID 16627130
- [Background] Raphael B, Wooding S, Stevens G, Connor J. Comorbidity: cannabis and complexity. J Psychiatr Pract. 2005 May;11(3):161-76. doi: 10.1097/00131746-200505000-00004. PMID 15920390
- [Background] Gilman SE, Abraham HD. A longitudinal study of the order of onset of alcohol dependence and major depression. Drug Alcohol Depend. 2001 Aug 1;63(3):277-86. doi: 10.1016/s0376-8716(00)00216-7. PMID 11418232
- [Background] Weisner C, Schmidt L. Gender disparities in treatment for alcohol problems. JAMA. 1992 Oct 14;268(14):1872-6. PMID 1328695
- [Background] Ananth J, Vandewater S, Kamal M, Brodsky A, Gamal R, Miller M. Missed diagnosis of substance abuse in psychiatric patients. Hosp Community Psychiatry. 1989 Mar;40(3):297-9. doi: 10.1176/ps.40.3.297. No abstract available. PMID 2917741
- [Background] Beckman LJ, Amaro H. Personal and social difficulties faced by women and men entering alcoholism treatment. J Stud Alcohol. 1986 Mar;47(2):135-45. doi: 10.15288/jsa.1986.47.135. PMID 3713175
- [Background] Babor TF, Higgins-Biddle JC. Alcohol screening and brief intervention: dissemination strategies for medical practice and public health. Addiction. 2000 May;95(5):677-86. doi: 10.1046/j.1360-0443.2000.9556773.x. PMID 10885042
- [Background] Whitlock EP, Polen MR, Green CA, Orleans T, Klein J; U.S. Preventive Services Task Force. Behavioral counseling interventions in primary care to reduce risky/harmful alcohol use by adults: a summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2004 Apr 6;140(7):557-68. doi: 10.7326/0003-4819-140-7-200404060-00017. PMID 15068985
- [Background] Institute of Medicine (US) Committee on Crossing the Quality Chasm: Adaptation to Mental Health and Addictive Disorders. Improving the Quality of Health Care for Mental and Substance-Use Conditions: Quality Chasm Series. Washington (DC): National Academies Press (US); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK19830/ PMID 20669433
- [Background] Mallin R, Slott K, Tumblin M, Hunter M. Detection of substance use disorders in patients presenting with depression. Subst Abus. 2002 Jun;23(2):115-20. doi: 10.1080/08897070209511481. PMID 12444356
- [Background] Gonzales JJ, Insel TR. The conundrum of co-occurring mental and substance use disorders: opportunities for research. Biol Psychiatry. 2004 Nov 15;56(10):723-5. doi: 10.1016/j.biopsych.2004.09.007. No abstract available. PMID 15556114
- [Background] Watkins KE, Burnam A, Kung FY, Paddock S. A national survey of care for persons with co-occurring mental and substance use disorders. Psychiatr Serv. 2001 Aug;52(8):1062-8. doi: 10.1176/appi.ps.52.8.1062. PMID 11474052
- [Background] Prochaska JJ, Fromont SC, Hall SM. How prepared are psychiatry residents for treating nicotine dependence? Acad Psychiatry. 2005 Jul-Aug;29(3):256-61. doi: 10.1176/appi.ap.29.3.256. PMID 16141120
- [Background] Sattar SP, Madison J, Markert RJ, Bhatia SC, Petty F. Addiction training scale: pilot study of a self-report evaluation tool for psychiatry residents. Acad Psychiatry. 2004 Fall;28(3):204-8. doi: 10.1176/appi.ap.28.3.204. PMID 15507555
- [Background] Renner JA Jr. How to train residents to identify and treat dual diagnosis patients. Biol Psychiatry. 2004 Nov 15;56(10):810-6. doi: 10.1016/j.biopsych.2004.04.003. PMID 15556127
- [Background] Mertens JR, Weisner C, Ray GT, Fireman B, Walsh K. Hazardous drinkers and drug users in HMO primary care: prevalence, medical conditions, and costs. Alcohol Clin Exp Res. 2005 Jun;29(6):989-98. doi: 10.1097/01.alc.0000167958.68586.3d. PMID 15976525
- [Background] Tiet QQ, Finney JW, Moos RH. Screening psychiatric patients for illicit drug use disorders and problems. Clin Psychol Rev. 2008 Apr;28(4):578-91. doi: 10.1016/j.cpr.2007.08.002. Epub 2007 Sep 8. PMID 17900773
- [Background] Cherpitel CJ, Ye Y. Drug use and problem drinking associated with primary care and emergency room utilization in the US general population: data from the 2005 national alcohol survey. Drug Alcohol Depend. 2008 Oct 1;97(3):226-30. doi: 10.1016/j.drugalcdep.2008.03.033. Epub 2008 May 21. PMID 18499355
- [Background] McGeary KA, French MT. Illicit drug use and emergency room utilization. Health Serv Res. 2000 Apr;35(1 Pt 1):153-69. PMID 10778828
- [Background] Kolbasovsky A, Futterman R. Predicting psychiatric emergency room recidivism. Manag Care Interface. 2007 Apr;20(4):33-8. PMID 17474328
- [Background] Prince JD, Akincigil A, Hoover DR, Walkup JT, Bilder S, Crystal S. Substance abuse and hospitalization for mood disorder among Medicaid beneficiaries. Am J Public Health. 2009 Jan;99(1):160-7. doi: 10.2105/AJPH.2007.133249. Epub 2008 Nov 13. PMID 19008505
- [Background] Cleary M, Hunt GE, Matheson S, Siegfried N, Walter G. Psychosocial treatment programs for people with both severe mental illness and substance misuse. Schizophr Bull. 2008 Mar;34(2):226-8. doi: 10.1093/schbul/sbm165. Epub 2008 Jan 29. PMID 18234699
- [Background] Partonen T, Sihvo S, Lonnqvist JK. Patients excluded from an antidepressant efficacy trial. J Clin Psychiatry. 1996 Dec;57(12):572-5. doi: 10.4088/jcp.v57n1203. PMID 9010119
- [Background] Posternak MA, Zimmerman M, Keitner GI, Miller IW. A reevaluation of the exclusion criteria used in antidepressant efficacy trials. Am J Psychiatry. 2002 Feb;159(2):191-200. doi: 10.1176/appi.ajp.159.2.191. PMID 11823258
- [Background] Sullivan PF, Joyce PR. Effects of exclusion criteria in depression treatment studies. J Affect Disord. 1994 Sep;32(1):21-6. doi: 10.1016/0165-0327(94)90057-4. PMID 7798463
- [Background] Havassy BE, Alvidrez J, Owen KK. Comparisons of patients with comorbid psychiatric and substance use disorders: implications for treatment and service delivery. Am J Psychiatry. 2004 Jan;161(1):139-45. doi: 10.1176/appi.ajp.161.1.139. PMID 14702262
- [Background] Volkow ND. The reality of comorbidity: depression and drug abuse. Biol Psychiatry. 2004 Nov 15;56(10):714-7. doi: 10.1016/j.biopsych.2004.07.007. No abstract available. PMID 15556111
- [Background] Compton WM 3rd, Cottler LB, Phelps DL, Ben Abdallah A, Spitznagel EL. Psychiatric disorders among drug dependent subjects: are they primary or secondary? Am J Addict. 2000 Spring;9(2):126-34. doi: 10.1080/10550490050173190. PMID 10934574
- [Background] Clark RE, Teague GB, Ricketts SK, Bush PW, Xie H, McGuire TG, Drake RE, McHugo GJ, Keller AM, Zubkoff M. Cost-effectiveness of assertive community treatment versus standard case management for persons with co-occurring severe mental illness and substance use disorders. Health Serv Res. 1998 Dec;33(5 Pt 1):1285-308. PMID 9865221
- [Background] Prochaska J, DiClemente C. Toward a comprehensive model of change. In: Miller W, Heather N, eds. Treating Addictive Behaviors: Processes of Change. New York: Plenum, 1984:3-27
- [Background] Miller WR, Rose GS. Toward a theory of motivational interviewing. Am Psychol. 2009 Sep;64(6):527-37. doi: 10.1037/a0016830. PMID 19739882
- [Background] Miller WR, Sanchez VC. Motivating young adults for treatment and lifestyle change. In: Howard GS, Nathan PE, eds. Alcohol Use and Misuse by Young Adults. Notra Dame, IN: University of Notre Dame Press, 1994:55-82
- [Background] Janis IL, Mann L. Decision Making : A Psychological Analysis of Conflict, Choice, and Commitment New York: Free Press, 1977
- [Background] Carey KB, Carey MP, Maisto SA, Henson JM. Brief motivational interventions for heavy college drinkers: A randomized controlled trial. J Consult Clin Psychol. 2006 Oct;74(5):943-54. doi: 10.1037/0022-006X.74.5.943. PMID 17032098
- [Background] Collins SE, Carey KB. Lack of effect for decisional balance as a brief motivational intervention for at-risk college drinkers. Addict Behav. 2005 Aug;30(7):1425-30. doi: 10.1016/j.addbeh.2005.01.004. PMID 16022936
- [Background] Wilk AI, Jensen NM, Havighurst TC. Meta-analysis of randomized control trials addressing brief interventions in heavy alcohol drinkers. J Gen Intern Med. 1997 May;12(5):274-83. doi: 10.1046/j.1525-1497.1997.012005274.x. PMID 9159696
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing People for Change. 2nd ed. New York: Guilford Press, 2002
- [Background] Moyers TB, Martin T, Manuel JK, Hendrickson SM, Miller WR. Assessing competence in the use of motivational interviewing. J Subst Abuse Treat. 2005 Jan;28(1):19-26. doi: 10.1016/j.jsat.2004.11.001. PMID 15723728
- [Background] McCambridge J, Strang J. The efficacy of single-session motivational interviewing in reducing drug consumption and perceptions of drug-related risk and harm among young people: results from a multi-site cluster randomized trial. Addiction. 2004 Jan;99(1):39-52. doi: 10.1111/j.1360-0443.2004.00564.x. PMID 14678061
- [Background] Martin G, Copeland J, Swift W. The Adolescent Cannabis Check-Up: feasibility of a brief intervention for young cannabis users. J Subst Abuse Treat. 2005 Oct;29(3):207-13. doi: 10.1016/j.jsat.2005.06.005. PMID 16183469
- [Background] Saunders B, Wilkinson C, Phillips M. The impact of a brief motivational intervention with opiate users attending a methadone programme. Addiction. 1995 Mar;90(3):415-24. doi: 10.1046/j.1360-0443.1995.90341510.x. PMID 7735025
- [Background] McCambridge J, Slym RL, Strang J. Randomized controlled trial of motivational interviewing compared with drug information and advice for early intervention among young cannabis users. Addiction. 2008 Nov;103(11):1809-18. doi: 10.1111/j.1360-0443.2008.02331.x. Epub 2008 Sep 4. PMID 18778385
- [Background] Otto C, Crackau B, Lohrmann I, Zahradnik A, Bischof G, John U, Rumpf HJ. Brief intervention in general hospital for problematic prescription drug use: 12-month outcome. Drug Alcohol Depend. 2009 Dec 1;105(3):221-6. doi: 10.1016/j.drugalcdep.2009.07.010. Epub 2009 Sep 1. PMID 19726140
- [Background] Wells-Parker E, Dill P, Williams M, Stoduto G. Are depressed drinking/driving offenders more receptive to brief intervention? Addict Behav. 2006 Feb;31(2):339-50. doi: 10.1016/j.addbeh.2005.05.011. Epub 2005 Jul 6. PMID 16005159
- [Background] Beich A, Thorsen T, Rollnick S. Screening in brief intervention trials targeting excessive drinkers in general practice: systematic review and meta-analysis. BMJ. 2003 Sep 6;327(7414):536-42. doi: 10.1136/bmj.327.7414.536. PMID 12958114
- [Background] Vasilaki EI, Hosier SG, Cox WM. The efficacy of motivational interviewing as a brief intervention for excessive drinking: a meta-analytic review. Alcohol Alcohol. 2006 May-Jun;41(3):328-35. doi: 10.1093/alcalc/agl016. Epub 2006 Mar 17. PMID 16547122
- [Background] Fleming M, Manwell LB. Brief intervention in primary care settings. A primary treatment method for at-risk, problem, and dependent drinkers. Alcohol Res Health. 1999;23(2):128-37. PMID 10890807
- [Background] Sellman JD, Sullivan PF, Dore GM, Adamson SJ, MacEwan I. A randomized controlled trial of motivational enhancement therapy (MET) for mild to moderate alcohol dependence. J Stud Alcohol. 2001 May;62(3):389-96. doi: 10.15288/jsa.2001.62.389. PMID 11414349
- [Background] Bertholet N, Daeppen JB, Wietlisbach V, Fleming M, Burnand B. Reduction of alcohol consumption by brief alcohol intervention in primary care: systematic review and meta-analysis. Arch Intern Med. 2005 May 9;165(9):986-95. doi: 10.1001/archinte.165.9.986. PMID 15883236
- [Background] Fleming MF, Mundt MP, French MT, Manwell LB, Stauffacher EA, Barry KL. Benefit-cost analysis of brief physician advice with problem drinkers in primary care settings. Med Care. 2000 Jan;38(1):7-18. doi: 10.1097/00005650-200001000-00003. PMID 10630716
- [Background] Fleming MF, Graham AW. Screening and brief interventions for alcohol use disorders in managed care settings. Recent Dev Alcohol. 2001;15:393-416. doi: 10.1007/978-0-306-47193-3_22. PMID 11449755
- [Background] Fleming MF, Mundt MP, French MT, Manwell LB, Stauffacher EA, Barry KL. Brief physician advice for problem drinkers: long-term efficacy and benefit-cost analysis. Alcohol Clin Exp Res. 2002 Jan;26(1):36-43. PMID 11821652
- [Background] Dinh-Zarr T, Diguiseppi C, Heitman E, Roberts I. Preventing injuries through interventions for problem drinking: a systematic review of randomized controlled trials. Alcohol Alcohol. 1999 Jul-Aug;34(4):609-21. doi: 10.1093/alcalc/34.4.609. PMID 10456590
- [Background] Saitz R, Svikis D, D'Onofrio G, Kraemer KL, Perl H. Challenges applying alcohol brief intervention in diverse practice settings: populations, outcomes, and costs. Alcohol Clin Exp Res. 2006 Feb;30(2):332-8. doi: 10.1111/j.1530-0277.2006.00038.x. PMID 16441282
- [Background] Grothues J, Bischof G, Reinhardt S, Hapke U, Meyer C, John U, Rumpf HJ. Intention to change drinking behaviour in general practice patients with problematic drinking and comorbid depression or anxiety. Alcohol Alcohol. 2005 Sep-Oct;40(5):394-400. doi: 10.1093/alcalc/agh182. Epub 2005 Jul 4. PMID 15996967
- [Background] Grothues JM, Bischof G, Reinhardt S, Meyer C, John U, Rumpf HJ. Effectiveness of brief alcohol interventions for general practice patients with problematic drinking behavior and comorbid anxiety or depressive disorders. Drug Alcohol Depend. 2008 Apr 1;94(1-3):214-20. doi: 10.1016/j.drugalcdep.2007.11.015. Epub 2008 Jan 22. PMID 18207336
- [Background] Kay-Lambkin FJ, Baker AL, Lewin TJ, Carr VJ. Computer-based psychological treatment for comorbid depression and problematic alcohol and/or cannabis use: a randomized controlled trial of clinical efficacy. Addiction. 2009 Mar;104(3):378-88. doi: 10.1111/j.1360-0443.2008.02444.x. PMID 19207345
- [Background] Baker A, Lewin T, Reichler H, Clancy R, Carr V, Garrett R, Sly K, Devir H, Terry M. Evaluation of a motivational interview for substance use within psychiatric in-patient services. Addiction. 2002 Oct;97(10):1329-37. doi: 10.1046/j.1360-0443.2002.00178.x. PMID 12359037
- [Background] Barrowclough C, Haddock G, Tarrier N, Lewis SW, Moring J, O'Brien R, Schofield N, McGovern J. Randomized controlled trial of motivational interviewing, cognitive behavior therapy, and family intervention for patients with comorbid schizophrenia and substance use disorders. Am J Psychiatry. 2001 Oct;158(10):1706-13. doi: 10.1176/appi.ajp.158.10.1706. PMID 11579006
- [Background] Graeber DA, Moyers TB, Griffith G, Guajardo E, Tonigan S. A pilot study comparing motivational interviewing and an educational intervention in patients with schizophrenia and alcohol use disorders. Community Ment Health J. 2003 Jun;39(3):189-202. doi: 10.1023/a:1023371705506. PMID 12836801
- [Background] Kavanagh DJ, Young R, White A, Saunders JB, Wallis J, Shockley N, Jenner L, Clair A. A brief motivational intervention for substance misuse in recent-onset psychosis. Drug Alcohol Rev. 2004 Jun;23(2):151-5. doi: 10.1080/09595230410001704127. PMID 15370020
- [Background] Martino S, Carroll KM, O'Malley SS, Rounsaville BJ. Motivational interviewing with psychiatrically ill substance abusing patients. Am J Addict. 2000 Winter;9(1):88-91. doi: 10.1080/10550490050172263. PMID 10914297
- [Background] Swanson AJ, Pantalon MV, Cohen KR. Motivational interviewing and treatment adherence among psychiatric and dually diagnosed patients. J Nerv Ment Dis. 1999 Oct;187(10):630-5. doi: 10.1097/00005053-199910000-00007. PMID 10535657
- [Background] Steinberg ML, Ziedonis DM, Krejci JA, Brandon TH. Motivational interviewing with personalized feedback: a brief intervention for motivating smokers with schizophrenia to seek treatment for tobacco dependence. J Consult Clin Psychol. 2004 Aug;72(4):723-8. doi: 10.1037/0022-006X.72.4.723. PMID 15301657
- [Background] Martino S, Carroll KM, Nich C, Rounsaville BJ. A randomized controlled pilot study of motivational interviewing for patients with psychotic and drug use disorders. Addiction. 2006 Oct;101(10):1479-92. doi: 10.1111/j.1360-0443.2006.01554.x. PMID 16968350
- [Background] Santa Ana EJ, Wulfert E, Nietert PJ. Efficacy of group motivational interviewing (GMI) for psychiatric inpatients with chemical dependence. J Consult Clin Psychol. 2007 Oct;75(5):816-22. doi: 10.1037/0022-006X.75.5.816. PMID 17907864
- [Background] Daley DC, Salloum IM, Zuckoff A, Kirisci L, Thase ME. Increasing treatment adherence among outpatients with depression and cocaine dependence: results of a pilot study. Am J Psychiatry. 1998 Nov;155(11):1611-3. doi: 10.1176/ajp.155.11.1611. PMID 9812129
- [Background] Joo JH, Solano FX, Mulsant BH, Reynolds CF, Lenze EJ. Predictors of adequacy of depression management in the primary care setting. Psychiatr Serv. 2005 Dec;56(12):1524-8. doi: 10.1176/appi.ps.56.12.1524. PMID 16339613
- [Background] Katon WJ. The Institute of Medicine "Chasm" report: implications for depression collaborative care models. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):222-9. doi: 10.1016/s0163-8343(03)00064-1. PMID 12850653
- [Background] Von Korff M, Katon W, Unutzer J, Wells K, Wagner EH. Improving depression care: barriers, solutions, and research needs. J Fam Pract. 2001 Jun;50(6):E1. PMID 11401751
- [Background] Blazer DG, Kessler RC, McGonagle KA, Swartz MS. The prevalence and distribution of major depression in a national community sample: the National Comorbidity Survey. Am J Psychiatry. 1994 Jul;151(7):979-86. doi: 10.1176/ajp.151.7.979. PMID 8010383
- [Background] Brown RA, Evans DM, Miller IW, Burgess ES, Mueller TI. Cognitive-behavioral treatment for depression in alcoholism. J Consult Clin Psychol. 1997 Oct;65(5):715-26. doi: 10.1037//0022-006x.65.5.715. PMID 9337490
- [Background] Hesse M. Achieving abstinence by treating depression in the presence of substance-use disorders. Addict Behav. 2004 Aug;29(6):1137-41. doi: 10.1016/j.addbeh.2004.03.006. PMID 15236814
- [Background] Humphreys K. Professional interventions that facilitate 12-step self-help group involvement. Alcohol Res Health. 1999;23(2):93-8. PMID 10890802
- [Background] Barry KL, (Consensus Panel Chair). Brief interventions and brief therapies for substance abuse. Treatment Improvement Protocol (TIP) Series 34. Rockville (MD): Substance Abuse and Mental Health Services Administration. DHHS Publication No. (SMA) 99-3353, 1999
- [Background] Morgenstern J, Bux DA Jr, Parsons J, Hagman BT, Wainberg M, Irwin T. Randomized trial to reduce club drug use and HIV risk behaviors among men who have sex with men. J Consult Clin Psychol. 2009 Aug;77(4):645-56. doi: 10.1037/a0015588. PMID 19634958
- [Background] Cutler RB, Fishbain DA. Are alcoholism treatments effective? The Project MATCH data. BMC Public Health. 2005 Jul 14;5:75. doi: 10.1186/1471-2458-5-75. PMID 16018798
- [Background] Arkowitz H, Westra HA. Introduction to the special series on motivational interviewing and psychotherapy. J Clin Psychol. 2009 Nov;65(11):1149-55. doi: 10.1002/jclp.20640. PMID 19785011
- [Background] Westra HA. Managing resistance in cognitive behavioural therapy: the application of motivational interviewing in mixed anxiety and depression. Cogn Behav Ther. 2004;33(4):161-75. doi: 10.1080/16506070410026426. PMID 15625790
- [Background] Galanter M. Innovations: alcohol & drug abuse: spirituality in Alcoholics Anonymous: a valuable adjunct to psychiatric services. Psychiatr Serv. 2006 Mar;57(3):307-9. doi: 10.1176/appi.ps.57.3.307. PMID 16524986
- [Background] Hansen LJ, Olivarius N, Beich A, Barfod S. Encouraging GPs to undertake screening and a brief intervention in order to reduce problem drinking: a randomized controlled trial. Fam Pract. 1999 Dec;16(6):551-7. doi: 10.1093/fampra/16.6.551. PMID 10625125
- [Background] McNally AM, Palfai TP, Kahler CW. Motivational interventions for heavy drinking college students: examining the role of discrepancy-related psychological processes. Psychol Addict Behav. 2005 Mar;19(1):79-87. doi: 10.1037/0893-164X.19.1.79. PMID 15783281
- [Background] Murphy JG, Correia CJ, Colby SM, Vuchinich RE. Using behavioral theories of choice to predict drinking outcomes following a brief intervention. Exp Clin Psychopharmacol. 2005 May;13(2):93-101. doi: 10.1037/1064-1297.13.2.93. PMID 15943542
- [Background] Mundt MP. Analyzing the costs and benefits of brief intervention. Alcohol Res Health. 2006;29(1):34-6. PMID 16767851
- [Background] Zarkin GA, Bray JW, Davis KL, Babor TF, Higgins-Biddle JC. The costs of screening and brief intervention for risky alcohol use. J Stud Alcohol. 2003 Nov;64(6):849-57. doi: 10.15288/jsa.2003.64.849. PMID 14743949
- [Background] Baer JS, Kivlahan DR, Blume AW, McKnight P, Marlatt GA. Brief intervention for heavy-drinking college students: 4-year follow-up and natural history. Am J Public Health. 2001 Aug;91(8):1310-6. doi: 10.2105/ajph.91.8.1310. PMID 11499124
- [Background] Nilssen O. Long-term effect of brief intervention in at-risk alcohol drinkers: a 9-year follow-up study. Alcohol Alcohol. 2004 Nov-Dec;39(6):548-51. doi: 10.1093/alcalc/agh095. Epub 2004 Sep 20. PMID 15381513
- [Background] Chi FW, Satre DD, Weisner C. Chemical dependency patients with cooccurring psychiatric diagnoses: service patterns and 1-year outcomes. Alcohol Clin Exp Res. 2006 May;30(5):851-9. doi: 10.1111/j.1530-0277.2006.00100.x. PMID 16634854
- [Background] Satre DD, Sterling SA, Mackin RS, Weisner C. Patterns of alcohol and drug use among depressed older adults seeking outpatient psychiatric services. Am J Geriatr Psychiatry. 2011 Aug;19(8):695-703. doi: 10.1097/JGP.0b013e3181f17f0a. PMID 21788921
- [Background] Mertens JR, Flisher AJ, Satre DD, Weisner CM. The role of medical conditions and primary care services in 5-year substance use outcomes among chemical dependency treatment patients. Drug Alcohol Depend. 2008 Nov 1;98(1-2):45-53. doi: 10.1016/j.drugalcdep.2008.04.007. Epub 2008 Jun 20. PMID 18571875
- [Background] Satre DD, Mertens J, Arean PA, Weisner C. Contrasting outcomes of older versus middle-aged and younger adult chemical dependency patients in a managed care program. J Stud Alcohol. 2003 Jul;64(4):520-30. doi: 10.15288/jsa.2003.64.520. PMID 12921194
- [Background] Satre DD, Knight BG, Dickson-Fuhrmann E, Jarvik LF. Substance abuse treatment initiation among older adults in the GET SMART program: effects of depression and cognitive status. Aging Ment Health. 2004 Jul;8(4):346-54. doi: 10.1080/13607860410001709692. PMID 15370050
- [Background] Satre DD, Mertens JR, Arean PA, Weisner C. Five-year alcohol and drug treatment outcomes of older adults versus middle-aged and younger adults in a managed care program. Addiction. 2004 Oct;99(10):1286-97. doi: 10.1111/j.1360-0443.2004.00831.x. PMID 15369567
- [Background] Satre DD, Gordon NP, Weisner C. Alcohol consumption, medical conditions, and health behavior in older adults. Am J Health Behav. 2007 May-Jun;31(3):238-48. doi: 10.5555/ajhb.2007.31.3.238. PMID 17402864
- [Background] Weisner C, Ray GT, Mertens JR, Satre DD, Moore C. Short-term alcohol and drug treatment outcomes predict long-term outcome. Drug Alcohol Depend. 2003 Sep 10;71(3):281-94. doi: 10.1016/s0376-8716(03)00167-4. PMID 12957346
- [Background] Satre DD, Kohn CS, Weisner C. Cigarette smoking and long-term alcohol and drug treatment outcomes: a telephone follow-up at five years. Am J Addict. 2007 Jan-Feb;16(1):32-7. doi: 10.1080/10550490601077825. PMID 17364419
- [Background] Weisner C, Lu Y, Hinman A, Monahan J, Bonnie RJ, Moore CD, Chi FW, Appelbaum PS. Substance use, symptom, and employment outcomes of persons with a workplace mandate for chemical dependency treatment. Psychiatr Serv. 2009 May;60(5):646-54. doi: 10.1176/ps.2009.60.5.646. PMID 19411353
- [Background] Satre DD, Arean PA. Effects of gender, ethnicity, and medical illness on drinking cessation in older primary care patients. J Aging Health. 2005 Feb;17(1):70-84. doi: 10.1177/0898264304272785. PMID 15601784
- [Background] Satre DD, Sterling S, Weisner C. Treatment of alcohol and drug problems in older women. Women in Recovery: Kaiser Permanente Women's Chemical Dependency Committee Newsletter. 2007;Winter:1-2
- [Background] Chi FW, Kaskutas LA, Sterling S, Campbell CI, Weisner C. Twelve-Step affiliation and 3-year substance use outcomes among adolescents: social support and religious service attendance as potential mediators. Addiction. 2009 Jun;104(6):927-39. doi: 10.1111/j.1360-0443.2009.02524.x. Epub 2009 Mar 13. PMID 19344442
- [Background] Chi FW, Weisner CM. Nine-year psychiatric trajectories and substance use outcomes: an application of the group-based modeling approach. Eval Rev. 2008 Feb;32(1):39-58. doi: 10.1177/0193841X07307317. PMID 18198170
- [Background] Satre DD, Blow FC, Chi FW, Weisner C. Gender differences in seven-year alcohol and drug treatment outcomes among older adults. Am J Addict. 2007 May-Jun;16(3):216-21. doi: 10.1080/10550490701375673. PMID 17612826
- [Background] Delucchi KL, Matzger H, Weisner C. Dependent and problem drinking over 5 years: a latent class growth analysis. Drug Alcohol Depend. 2004 Jun 11;74(3):235-44. doi: 10.1016/j.drugalcdep.2003.12.014. PMID 15194201
- [Background] Delucchi KL, Matzger H, Weisner C. Alcohol in emerging adulthood: 7-year study of problem and dependent drinkers. Addict Behav. 2008 Jan;33(1):134-42. doi: 10.1016/j.addbeh.2007.04.027. Epub 2007 May 3. PMID 17537582
- [Background] Parthasarathy S, Mertens J, Moore C, Weisner C. Utilization and cost impact of integrating substance abuse treatment and primary care. Med Care. 2003 Mar;41(3):357-67. doi: 10.1097/01.MLR.0000053018.20700.56. PMID 12618639
- [Background] Parthasarathy S, Weisner CM. Five-year trajectories of health care utilization and cost in a drug and alcohol treatment sample. Drug Alcohol Depend. 2005 Nov 1;80(2):231-40. doi: 10.1016/j.drugalcdep.2005.04.004. PMID 15916868
- [Background] Paperny DM, Aono JY, Lehman RM, Hammar SL, Risser J. Computer-assisted detection and intervention in adolescent high-risk health behaviors. J Pediatr. 1990 Mar;116(3):456-62. doi: 10.1016/s0022-3476(05)82844-6. PMID 2308041
- [Background] Chi FW, Sterling S, Weisner C. Adolescents with co-occurring substance use and mental conditions in a private managed care health plan: prevalence, patient characteristics, and treatment initiation and engagement. Am J Addict. 2006;15 Suppl 1:67-79. doi: 10.1080/10550490601006022. PMID 17182422
- [Background] Chi F, Weisner C. Continuity of care and costs among patients dually diagnosed with substance use disorders and parity psychiatric conditions in private managed care. Addiction Health Services Research Conference, Santa Monica, CA, Oct 25, 2005
- [Background] McLellan AT, Alterman AI, Metzger DS, Grissom GR, Woody GE, Luborsky L, O'Brien CP. Similarity of outcome predictors across opiate, cocaine, and alcohol treatments: role of treatment services. J Consult Clin Psychol. 1994 Dec;62(6):1141-58. doi: 10.1037//0022-006x.62.6.1141. PMID 7860812
- [Background] Mohr DC, Hart SL, Julian L, Catledge C, Honos-Webb L, Vella L, Tasch ET. Telephone-administered psychotherapy for depression. Arch Gen Psychiatry. 2005 Sep;62(9):1007-14. doi: 10.1001/archpsyc.62.9.1007. PMID 16143732
- [Background] Keller MB, Hanks DL. Anxiety symptom relief in depression treatment outcomes. J Clin Psychiatry. 1995;56 Suppl 6:22-9. PMID 7649969
- [Background] Kessler RC, Gruber M, Hettema JM, Hwang I, Sampson N, Yonkers KA. Co-morbid major depression and generalized anxiety disorders in the National Comorbidity Survey follow-up. Psychol Med. 2008 Mar;38(3):365-74. doi: 10.1017/S0033291707002012. Epub 2007 Nov 30. PMID 18047766
- [Background] Levin FR, Hennessy G. Bipolar disorder and substance abuse. Biol Psychiatry. 2004 Nov 15;56(10):738-48. doi: 10.1016/j.biopsych.2004.05.008. PMID 15556118
- [Background] Herzog DB, Franko DL, Dorer DJ, Keel PK, Jackson S, Manzo MP. Drug abuse in women with eating disorders. Int J Eat Disord. 2006 Jul;39(5):364-8. doi: 10.1002/eat.20257. PMID 16565976
- [Background] Franko DL, Dorer DJ, Keel PK, Jackson S, Manzo MP, Herzog DB. Interactions between eating disorders and drug abuse. J Nerv Ment Dis. 2008 Jul;196(7):556-61. doi: 10.1097/NMD.0b013e31817d0153. PMID 18626296
- [Background] Westermeyer J. Comorbid schizophrenia and substance abuse: a review of epidemiology and course. Am J Addict. 2006 Sep-Oct;15(5):345-55. doi: 10.1080/10550490600860114. PMID 16966190
- [Background] Green AI, Brown ES. Comorbid schizophrenia and substance abuse. J Clin Psychiatry. 2006 Sep;67(9):e08. PMID 17081075
- [Background] Kaiser Permanente Northern California Dual Diagnosis Best Practices Committee. Recommendations for Improving Treatment of Co-Occurring Disorders. Oakland, Ca: Kaiser Permanente Medical Care Program; Sep 2007
- [Background] Kaiser Permanente Care Management Institute. Depression clinical practice guidelines. http://www.guideline.gov/summary/summary.aspx?doc_id=9632&nbr=005152&string=kaiser. Published 2006. Accessed Jan 9, 2009
- [Background] Beck AT, Rush AJ, Shaw BF, et al. Cognitive Therapy of Depression. New York: Guildford Press, 1979
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Stahl SM. Selecting an antidepressant by using mechanism of action to enhance efficacy and avoid side effects. J Clin Psychiatry. 1998;59 Suppl 18:23-9. PMID 9840195
- [Background] Flanagan RJ. Fatal toxicity of drugs used in psychiatry. Hum Psychopharmacol. 2008 Jan;23 Suppl 1:43-51. doi: 10.1002/hup.916. PMID 18098225
- [Background] Horgan CM, Merrick EL, Stewart MT, Scholle SH, Shih S. Improving medication management of depression in health plans. Psychiatr Serv. 2008 Jan;59(1):72-7. doi: 10.1176/ps.2008.59.1.72. PMID 18182542
- [Background] Sobell LC, Sobell MB. Alcohol Consumption Measures. In: Allen JP, Wilson VB, eds. Assessing Alcohol Problems. A Guide for Clinicians and Researchers. 2nd ed. Bethesda, MD: National Institute on Alcohol Abuse and Alcoholism, 2003:75-100
- [Background] Del Boca FK, Darkes J. The validity of self-reports of alcohol consumption: state of the science and challenges for research. Addiction. 2003 Dec;98 Suppl 2:1-12. doi: 10.1046/j.1359-6357.2003.00586.x. PMID 14984237
- [Background] Chermack ST, Singer K, Beresford TP. Screening for alcoholism among medical inpatients: how important is corroboration of patient self-report? Alcohol Clin Exp Res. 1998 Oct;22(7):1393-8. doi: 10.1111/j.1530-0277.1998.tb03925.x. PMID 9802518
- [Background] Midanik LT. Validity of self-reported alcohol use: a literature review and assessment. Br J Addict. 1988 Sep;83(9):1019-30. doi: 10.1111/j.1360-0443.1988.tb00526.x. No abstract available. PMID 3066418
- [Background] O'Farrell TJ, Fals-Stewart W, Murphy M. Concurrent validity of a brief self-report Drug Use Frequency measure. Addict Behav. 2003 Mar;28(2):327-37. doi: 10.1016/s0306-4603(01)00226-x. PMID 12573682
- [Background] Sohn MW, Zhang H, Arnold N, Stroupe K, Taylor BC, Wilt TJ, Hynes DM. Transition to the new race/ethnicity data collection standards in the Department of Veterans Affairs. Popul Health Metr. 2006 Jul 6;4:7. doi: 10.1186/1478-7954-4-7. PMID 16824220
- [Background] National Institute on Drug Abuse. Screening for tobacco, alcohol and other drug use. http://www.drugabuse.gov/nidamed/screening/. Published 2009. Updated Sep 22, 2009. Accessed Oct 9, 2009
- [Background] Humeniuk R, Ali R, Babor TF, Farrell M, Formigoni ML, Jittiwutikarn J, de Lacerda RB, Ling W, Marsden J, Monteiro M, Nhiwatiwa S, Pal H, Poznyak V, Simon S. Validation of the Alcohol, Smoking And Substance Involvement Screening Test (ASSIST). Addiction. 2008 Jun;103(6):1039-47. doi: 10.1111/j.1360-0443.2007.02114.x. Epub 2008 Mar 28. PMID 18373724